CLINICAL TRIAL: NCT02057341
Title: A Study of ARRY-371797 in Patients With LMNA-Related Dilated Cardiomyopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARRAY-797-231; C4411004 (Other: Pfizer)
Record Dates: First submitted 2014-02-05; First posted 2014-02-07 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: LMNA-Related Dilated Cardiomyopathy
Keywords: laminopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated; Laminopathies | interventions — ARRY-371797

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ARRY-371797 (Dose 1) (Experimental)
  Interventions: Drug: ARRY-371797, p38 inhibitor; oral
- ARRY-371797 (Dose 2) (Experimental)
  Interventions: Drug: ARRY-371797, p38 inhibitor; oral

INTERVENTIONS:
Drug: ARRY-371797, p38 inhibitor; oral — multiple dose, single schedule

SUMMARY:
This is a Phase 2 pilot study, involving a 48-week treatment period, designed to test the effectiveness of investigational study drug ARRY-371797 in treating patients with symptomatic genetic dilated cardiomyopathy due to a lamin A/C gene mutation, and to further evaluate the drug's safety. Approximately 12 patients from the US will be enrolled in this study.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients with idiopathic dilated cardiomyopathy and stable New York Heart Association (NYHA) Class II - IIIa congestive heart failure (CHF).
* Stable, guidelines-based medical and device therapy, without any CHF hospitalizations or change in heart failure drug dose with ≥ 50% reduction in dose or ≥ 100% increase in dose in the past 3 months.
* Left ventricular (LV) end diastolic diameter by trans-thoracic echocardiography of > 3.3 cm/m2 (for females) or 3.4 cm/m2 (for males) and/or LV ejection fraction ≤ 45%.
* Gene positive for a pathogenic mutation in the LMNA gene, as determined by a CLIA-certified clinical laboratory (mutations including but not limited to: splice-site, non-sense, deletion mutations, a mis-sense mutation in a highly conserved codon, a mis-sense mutation involving a major charge change, a mis-sense mutation previously associated with genetic dilated cardiomyopathy).
* Within 3 weeks prior to first dose of study drug, completed distance during six minute walk test of ≥ 100 m and ≤ 350 m AND/OR ≥ 100 m and ≤ 450 m AND ≤ 60% predicted distance AND patient is symptomatic for dilated cardiomyopathy per Investigator judgment.
* On the day before and day of first dose of study drug, completed distance during six minute walk test of ≥ 100 m and ≤ 400 m (with the greater value within 10% of the lesser value) AND/OR ≥ 100 m and ≤ 475 m (with the greater value within 10% of the lesser value) AND patient is symptomatic for dilated cardiomyopathy per Investigator judgment.
* Acceptable hematology, hepatic and renal function laboratory values within 3 weeks prior to first dose of study drug.
* Additional criteria exist.

Key Exclusion Criteria:

* Unstable clinical cardiac symptoms requiring unscheduled hospitalization within 60 days prior to study start.
* Clinically significant coronary artery disease, as per Investigator judgment.
* Currently receiving continuous intravenous (IV) inotrope infusion, or presence of a ventricular assist device, or history of prior heart transplantation.
* Any of the following within 60 days prior to study start: Myocardial infarction, cardiac surgical procedures, acute coronary syndrome, hemodynamically destabilizing cardiac arrhythmia, serious systemic infection with evidence of septicemia, any major surgical procedure requiring general anesthesia.
* Uncorrected, hemodynamically significant primary valvular disease.
* Initiation of cardiac resynchronization therapy within 180 days prior to study start.
* Likelihood, in the Investigator's opinion, of undergoing cardiac transplantation, left ventricular assist device or other device implantation, or other cardiac surgery within the next 6 months; or of requiring continuous IV inotropic treatment, or referral for hospice or end-of-life treatment.
* Active malignancy (except surgically-curative basal cell carcinoma, squamous cell carcinoma, or cervical carcinoma).
* Receiving chronic immunosuppressant therapy.
* Known positive serology for the human immunodeficiency virus (HIV), active hepatitis B and/or hepatitis C.
* Participation in any other investigational study of drugs or devices within 30 days prior to study start.
* Additional criteria exist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Assess the efficacy of the study drug in terms of change from Baseline in 6-minute walk test. | 12 weeks

SECONDARY OUTCOMES:
Assess the efficacy of study drug in terms of left ventricular function. | 48 weeks
Assess the efficacy of study drug in terms of right ventricular function. | 48 weeks
Assess the safety of study drug in terms of adverse events, clinical laboratory tests and electrocardiograms. | 48 weeks
Characterize the pharmacokinetics (PK) of study drug and metabolites in terms of plasma concentration-time profiles and model-based PK parameters. | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- United States (6):
  - Stanford University School of Medicine, Stanford, California
  - University of Colorado School of Medicine, Aurora, Colorado
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - The Ohio State University, Columbus, Ohio
  - Meriter Wisconsin Heart, Madison, Wisconsin

REFERENCES:
- [Derived] Garcia-Pavia P, Palomares JFR, Sinagra G, Barriales-Villa R, Lakdawala NK, Gottlieb RL, Goldberg RI, Elliott P, Lee P, Li H, Angeli FS, Judge DP, MacRae CA; REALM-DCM Investigators. REALM-DCM: A Phase 3, Multinational, Randomized, Placebo-Controlled Trial of ARRY-371797 in Patients With Symptomatic LMNA-Related Dilated Cardiomyopathy. Circ Heart Fail. 2024 Jul;17(7):e011548. doi: 10.1161/CIRCHEARTFAILURE.123.011548. Epub 2024 Jul 9. PMID 38979608
- [Derived] Judge DP, Taylor MR, Li H, Oliver C, Angeli FS, Lee PA, MacRae CA. Long-term effectiveness of ARRY-371797 in people with dilated cardiomyopathy and a faulty LMNA gene: a plain language summary. Future Cardiol. 2023 Mar;19(3):117-126. doi: 10.2217/fca-2022-0125. Epub 2023 Apr 3. PMID 37010012
- [Derived] MacRae CA, Taylor MR, Mestroni L, Moses J, Ashley EA, Wheeler MT, Lakdawala NK, Hershberger RE, Sandor V, Saunders ME, Oliver C, Lee PA, Judge DP. Plain Language Summary of Publication of the safety and efficacy of ARRY-371797 in people with dilated cardiomyopathy and a faulty LMNA gene. Future Cardiol. 2023 Feb;19(2):55-63. doi: 10.2217/fca-2022-0099. Epub 2023 Jan 31. PMID 36718638
- [Derived] MacRae CA, Taylor MRG, Mestroni L, Moses J, Ashley EA, Wheeler MT, Lakdawala NK, Hershberger RE, Sandor V, Saunders ME, Oliver C, Lee PA, Judge DP. Efficacy and Safety of ARRY-371797 in LMNA-Related Dilated Cardiomyopathy: A Phase 2 Study. Circ Genom Precis Med. 2023 Feb;16(1):e003730. doi: 10.1161/CIRCGEN.122.003730. Epub 2022 Dec 14. PMID 36515663